CLINICAL TRIAL: NCT06640439
Title: LED Therapy Using 830 Nm in the Mandibular Third Molar Surgery: Double-blind Randomized Clinical Trial.
Brief Title: LED Therapy for Third Molar Surgery
Acronym: LTTMS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yanjun Dan, Medical Doctor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2024-1088; Self-financed (Other: Self-financed)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Molar, Third; Photobiomodulation; Photobiomodulation Therapy; Third Molar Surgery
Keywords: photobiomodulation; LED; 830 nm; third molar surgery
MeSH Terms: interventions — Low-Level Light Therapy; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Patients who underwent mandibular third molar extraction
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study was a double-blind study in which the patient, the surgeon, and the statistician were all unaware of whether the patient received treatment or a placebo control light . Only the operator using the LED light was aware of this information. The assigned group was recorded on sealed and opaque envelopes. These cards were prepared by an independent person who was not involved in the study protocol. Once the patient underwent extraction and agreed to participate in this trial, this independent person opened the envelope to reveal the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Sham Comparator): The irradiation protocol was the same as that of the experimental group, and the light source used was simulated light. After surgery, patients took ibuprofen 0.3 g bid for 3 consecutive days, metronidazole 0.1 g tid, and cefaclor 0.375 g bid for 7 consecutive days.
  Interventions: Drug: Antibiotic
- Treatment Group (Experimental): LED light was irradiated 4 times (830 nm, 50 mW/cm2, 60 J/cm2, 1200 s) on D1 (before and after surgery), D2, and D3, which was extraoral irradiation. After surgery, ibuprofen 0.3 g bid for 3 consecutive days, metronidazole 0.1 g tid, and cefaclor 0.375 g bid for 7 consecutive days were taken.
  Interventions: Device: photobiomodulation; Drug: Antibiotic

INTERVENTIONS:
Device: photobiomodulation — 830 nm LED was used to irradiate the post-extraction area
  Arms: Treatment Group
Drug: Antibiotic — ibuprofen 0.3 g bid for 3 days, metronidazole 0.1 g tid, and cefaclor 0.375 g bid for 7 days after surgery

SUMMARY:
LED Therapy for third molar surgery

DETAILED DESCRIPTION:
LED Therapy using 830 nm in the mandibular third molar surgery

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Asians;
2. 20-55 years old;
3. Having mandibular third molars that are inappropriately erupted and need to be extracted due to caries, orthodontic reasons and/or periodontal disease;

Exclusion Criteria:

1. Underlying diseases: diabetes, cardiovascular disease, coagulation disorder, osteoporosis, hypertension, neurological disease, psychological disorder, tumor, systemic infection or cyst at the extraction site;
2. Women who are preparing for pregnancy, pregnant or breastfeeding;
3. Medication history: use of analgesics, anti-inflammatory drugs and/or antibacterial drugs 2 weeks before tooth extraction, need for systemic medication other than acetaminophen after surgery, allergy to acetaminophen, use of anticoagulants, bisphosphonates;
4. Bad habits, such as addicted to smoking, drinking, etc.;
5. Volunteers who have recently participated in other clinical trials;

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Pain | Day 7
  Visual Analogue Scale，VAS
Swelling | Day 3; Day 7
  Facial swelling was measured in 2 planes: the distance between the tragus and lip commissure and the distance between the gonion and external canthus of the eye.
Trismus | Day 3; Day 7
  Trismus was evaluated by measuring the maximum mouth opening between the edges of the upper and lower central incisors with a calibrated ruler.

SECONDARY OUTCOMES:
Quality of life score | Day 3; Day 7
  OHIP-14 Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided